CLINICAL TRIAL: NCT00973180
Title: Enhanced Prescription Drug Label to Improve Patient Understanding and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NU-0923017
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Prescription Medication Understanding
Keywords: Prescription medication understanding among diabetic and hypertension patients.; Prescription medication use among diabetic and hypertension patients.; Hemoglobin A1c changes among diabetic patients.; Blood pressure changes among hypertension patients.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Label (Experimental): Subjects in this arm will receive their prescriptions labeled with our enhanced, patient-friendly label.
  Interventions: Other: Enhanced Label
- Standard Label (No Intervention): Subjects in this arm will receive their prescriptions labeled with a standard label.

INTERVENTIONS:
Other: Enhanced Label — A prescription drug label that has simplified text, more white space and overall is more patient-friendly.
  Arms: Enhanced Label

SUMMARY:
The overall objective of this study is to test the efficacy of an evidence-based, enhanced Rx container label design to improve patients' understanding of instructions for use.

The investigators will conduct a randomized controlled trial (N=960) to evaluate the efficacy of the enhanced Rx container label to improve patients' understanding of actual prescribed medicines, compared to a standard label format. Patients with type II diabetes and/or hypertension at safety-net clinics affiliated with one central-fill pharmacy (Nova Scripts Central - NSC) receive their prescribed medicines from this location. Recruited subjects in this study will be randomly assigned to either intervention (enhanced Rx container label) or control (standard Rx label). All pill-form, regular dosing schedule medicines, including diabetes and hypertensive (i.e. ACE inhibitor) medicines associated with patients' treatment will be labeled according to study arm by the central-fill pharmacy. Study subjects will be interviewed at the time of dispensing the prescribed medicines at the clinic, again three months later (dispensing of refill), and finally nine months after baseline (dispensing of refill). Pharmacy refill data and medical record information - linked at these clinics - will be collected for exploratory analyses. Patients' ability to read and demonstrate Rx label instructions, including auxiliary warnings, will be the primary outcomes. Other exploratory outcome measures will also be measured, including 1) adverse effects associated with medication use defined by a) the rate of physician visits, b) the rate of emergency room visits, and c) the rate of hospitalizations and hospital admissions via emergency rooms for medication side effects (e.g. hyperglycemia or hypoglycemia); and 2) health outcome as measured by the change from baseline in hemoglobin A1c (HbA1c) and blood pressure measurements. Data from the actual use trial will be processed, reviewed, analyzed (in order of hypotheses), and reports prepared during the final months of this last phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type II diabetes or hypertension in their medical chart.
* 30 years or older.
* Fluent in English.

Exclusion Criteria:

* Uncorrectable hearing or visual impairment.
* Too ill to participate.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Understanding of prescription medication | Baseline, 3 months, 9 months

SECONDARY OUTCOMES:
Change in HbA1c or blood pressure readings | Baseline, 3 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Wolf, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wolf MS, Davis TC, Curtis LM, Bailey SC, Knox JP, Bergeron A, Abbet M, Shrank WH, Parker RM, Wood AJ. A Patient-Centered Prescription Drug Label to Promote Appropriate Medication Use and Adherence. J Gen Intern Med. 2016 Dec;31(12):1482-1489. doi: 10.1007/s11606-016-3816-x. Epub 2016 Aug 19. PMID 27542666